CLINICAL TRIAL: NCT05306548
Title: The NOR-CACTUS Trial - A Norwegian Trial Comparing Treatment Strategies for Carpal Tunnel Syndrome
Brief Title: A Norwegian Trial Comparing Treatment Strategies for Carpal Tunnel Syndrome
Acronym: NOR-CACTUS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Oslo University Hospital (Other); Vestre Viken Hospital Trust (Other); South-Eastern Norway Regional Health Authority (Other); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Hilde Berner Hammer, Principal Investigator, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIA2021-8
Record Dates: First submitted 2022-03-14; First posted 2022-04-01 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Surgery; Corticosteroid injection; Ultrasound guided intervention; Nerve conduction studies; Randomized controlled trial
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Injections; triamcinolone hexacetonide

STUDY DESIGN:
Intervention Model Description: Two-arm, prospective, multi-center, parallel-group, open-label assessor-blinded non-inferiority treatment strategy study
Who Masked: Outcomes Assessor
Masking Description: Participants in both strategy arms will have the site for injection/surgery covered with a adhesive bandage prior to assessment by blinded outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surgery treatment strategy (Active Comparator): Primary open surgical carpal tunnel release. Treatment effect is monitored on scheduled follow-up visits. Re-operation may be performed if medically indicated (e.g. postoperative complication, or failure of the primary procedure)
  Interventions: Procedure: Surgical carpal tunnel release
- Injection treatment strategy (Experimental): Primary treatment with ultrasound-guided corticosteroid injection. Treatment effect is monitored on scheduled follow-up visits. One additional injection may be administered, and subsequently surgical carpal tunnel release is performed in case of unsatisfactory treatment effect of the injection therapy. Treatment effect is graded on a 5-leve scale by subject from 1 (complete improvement) to 5 (severe worsening) of symptoms. Incomplete improvement (score 2 or higher) results in a second injection or secondary surgery.
  Interventions: Procedure: Surgical carpal tunnel release; Drug: Injection, Triamcinolone Hexacetonide, Per 5 Mg

INTERVENTIONS:
Procedure: Surgical carpal tunnel release — Open surgical division of the flexor retinaculum of the palm/wrist to release pressure on the median nerve
  Other Names: Open surgical carpal tunnel release
Drug: Injection, Triamcinolone Hexacetonide, Per 5 Mg — Ultrasound-guided injection of 20 mg of triamcinolone hexacetonide (or -acetonide) into the carpal tunnel space close to the median nerve
  Other Names: Ultrasound-guided corticosteroid injection
  Arms: Injection treatment strategy

SUMMARY:
Carpal tunnel syndrome (CTS) causes numbness and pain in the hand and arm, and is an important cause of work absence and disability. The aim of the NOR-CACTUS Trial is to compare outcomes of a treatment strategy where the initial treatment is up to two ultrasound-guided corticosteroid injections, followed by scheduled clinical assessment of treatment effect, and subsequent surgery if needed, to a treatment strategy where surgery is the first-line treatment. Participants will be randomized to one of the treatment strategies, and followed up for two years after start of the study intervention. Outcomes will include patient-reported, clinical, functional and neurophysiological measures, and health-economic aspects. The hypothesis of the study is that there is no difference between the two treatment groups in the percentage of patients with a satisfactory symptom relief (treatment success) one year after the initial therapeutic intervention.

DETAILED DESCRIPTION:
CTS is the most common non-traumatic hand disorder, prevalent in approximately 4% of the adult population. The condition may have a substantial impact on an individual's quality of life, ability to accomplish activities of daily living, and to perform occupational duties. Associated healthcare costs represent a significant socioeconomic burden.

Currently, many patients with mild and moderate CTS treated surgically without a preceding trial of less invasive non-surgical therapies. An increase in the use of non-surgical first-line therapies (e.g. corticosteroid injection into the carpal tunnel), while reserving surgery for refractory cases, aim to optimize the trade-off between treatment risk and benefit, while also ensuring appropriate use of health resources. However, there is a lack of studies directly comparing the efficacy of corticosteroid injections to surgery, and the long-term safety of corticosteroid injections has not been investigated.

It is not well-known if patients who are initially treated with corticosteroid injections will eventually need to proceed to surgery, and therefore may have to endure the symptoms for a longer period of time, with potentially worse long-term outcomes, compared to patients who has surgery as first-line treatment. On the other hand, it is not beneficial if patients are unnecessarily exposed to the risks associated with surgery, if symptoms could have been satisfactory resolved with a non-surgical method.

The current study will assess if first-line treatment with up to two ultrasound-guided corticosteroid injections is non-inferior to surgery with regards to treatment success. A less invasive treatment approach might result in important benefits to the patient, e.g. less pain, reduced risk of complications, and faster return to work and activities. This might also be of importance to family members, as many CTS patients are at an age where they have care responsibilities. Non-surgical treatments might benefit society by decreasing work absence and reducing health expenditure, and allowing better access to surgical services for other patient groups. High quality documentation is needed to provide a base for future treatment guidelines. Evidence based clinical guidelines provide treatment decision support and help reduce national and regional differences in treatment practices, and ensure that all patients have equal access to evidence-based treatment.

In the NOR-CACTUS trial, adult individuals with idiopathic CTS of a mild-to-moderate degree will be randomized to receive either A) Primary open surgical carpal tunnel release, or B) Up to two ultrasound-guided corticosteroid (triamcinolone hexacetonide) injections in the carpal tunnel, and subsequent open surgical carpal tunnel release in case of unsatisfactory treatment result. Participants will be randomized to receive one of the treatment strategies, and followed for two years, with the primary endpoint being successful treatment result one year after start of the intervention.

The hypothesis of the study is that the percentage of patients with a satisfactory symptom relief (treatment success) one year after the initial therapeutic intervention in the injection treatment strategy arm is non-inferior to that of the surgery treatment arm. The primary outcome is based on the disease-specific patient-reported outcome Boston Carpal Tunnel Questionnaire (BCTQ) symptom severity scale (SSS). Further outcomes will include other patient-reported, clinical, functional and neurophysiological measures, and health-economic aspects.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years of age)
2. Patient history indicating CTS
3. Neurophysiological examination performed within 6 months
4. Diagnosis of CTS based on:

   1. Classic/probable or possible symptoms, and neurophysiological findings consistent with CTS

      Or, in case of normal neurophysiological findings:
   2. Classic/probable symptoms and positive physical exam findings and/or nighttime symptoms
5. Mild to moderate symptoms (intermittent, interfering with everyday life, and/or disturb sleep)

Exclusion Criteria:

1. Previous CTS surgery or corticosteroid injection in the carpal tunnel in the relevant hand
2. Diagnosis of severe CTS, based on history and examination indicating severe CTS with constant symptoms including pain, loss of sensibility, dexterity or reduced temperature sensation, weakness of thumb abduction and opposition, or atrophy of thenar musculature. Disappearance of pain may indicate permanent sensory loss.
3. History suggesting underlying causes of CTS e.g. inflammatory wrist arthritis and/or flexor tenosynovitis
4. Previous significant trauma or fracture, deformity or tumor in the wrist or hand in the relevant hand
5. Presence of conditions affecting a normal nerve function e.g. cervical disc herniation, polyneuropathy or previous nerve injury
6. Major co-morbidities, such as severe malignancies, severe or uncontrolled infections, uncontrollable hypertension, severe cardiovascular disease (NYHA class III or IV) and/or severe respiratory diseases, severe renal failure, active ulcus ventriculi, leukopenia and/or thrombocytopenia
7. Severe psychiatric or mental disorders
8. Local infection or wound in the affected hand/wrist
9. Any other medical condition that according to the treating physician and/or local guidelines makes adherence to treatment protocol impossible
10. Inadequate birth control1, pregnancy2, and/or breastfeeding (current at screening or planned within the duration of the study)
11. Known hypersensitivity to Triamcinolone Hexacetonide (Lederspan) or any of the excipients (sorbitol, polysorbate or benzyl alcohol)
12. Concomitant therapy with CYP3A-inhibitors or digitalis glycosides
13. Patients vaccinated or immunized with live virus vaccines within 2 weeks of treatment
14. Alcohol or other substance abuse
15. Language barriers
16. Other factors which make adherence to study protocol impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Successful treatment result after 12 months | 12 months
  Boston Carpal Tunnel Questionnaire Symptom Severity Scale ≤ 1.5 after 12 months
  Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ SSS, Levine et. al 1993) is a disease-specific patient-reported outcome for CTS-related symptom severity. 11 items are scored by the patient on an ordinal scale from 1 (best) to 5 (worst), providing a mean score ranged 1-5. The primary outcome measure is achievement of BCTQ SSS ≤ 1.5, interpreted as a successful treatment result, 12 months after start of the study intervention.

SECONDARY OUTCOMES:
Successful treatment result after 3 months | 3 months
  Boston Carpal Tunnel Questionnaire Symptom Severity Scale ≤ 1.5 after 3 months
  Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ SSS, Levine et. al 1993) is a disease-specific patient-reported outcome for CTS-related symptom severity. 11 items are scored by the patient on an ordinal scale from 1 (best) to 5 (worst), providing a mean score ranged 1-5. The outcome measure is achievement of BCTQ SSS ≤ 1.5, interpreted as a successful treatment result, 3 months after start of the study intervention.
Successful treatment result after 6 months | 6 months
  Boston Carpal Tunnel Questionnaire Symptom Severity Scale ≤ 1.5 after 6 months
  Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ SSS, Levine et. al 1993) is a disease-specific patient-reported outcome for CTS-related symptom severity. 11 items are scored by the patient on an ordinal scale from 1 (best) to 5 (worst), providing a mean score ranged 1-5. The outcome measure is achievement of BCTQ SSS ≤ 1.5, interpreted as a successful treatment result, 6 months after start of the study intervention.
Successful treatment result after 24 months | 24 months
  Boston Carpal Tunnel Questionnaire Symptom Severity Scale ≤ 1.5 after 24 months
  Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ SSS, Levine et. al 1993) is a disease-specific patient-reported outcome for CTS-related symptom severity. 11 items are scored by the patient on an ordinal scale from 1 (best) to 5 (worst), providing a mean score ranged 1-5. The outcome measure is achievement of BCTQ SSS ≤ 1.5, interpreted as a successful treatment result, 24 months after start of the study intervention.
Boston Carpal Tunnel Questionnaire Symptom Severity Scale | 0-24 months
  Boston Carpal Tunnel Questionnaire Symptom Severity Scale (range 1-5)
  Boston Carpal Tunnel Questionnaire Symptom Severity Scale (BCTQ SSS, Levine et. al 1993) is a disease-specific patient-reported outcome for CTS-related symptom severity. 11 items are scored by the patient on an ordinal scale from 1 (best) to 5 (worst), providing a mean score ranged 1-5, used as outcome measure.
Boston Carpal Tunnel Questionnaire Functional Status Scale | 0-24 months
  Boston Carpal Tunnel Questionnaire Functional Status Scale (range 1-5)
  Boston Carpal Tunnel Questionnaire Functional Status Scale (BCTQ FSS, Levine et. al 1993) is a disease-specific patient-reported outcome for CTS-related functional impairment. 11 items are scored by the patient on an ordinal scale from 1 (best) to 5 (worst), providing a mean score ranged 1-5, used as outcome measure.
Nerve conduction studies: Motor median nerve distal latency | 0 and 12 months
  Nerve conduction studies of motor median nerve distal latency (milliseconds)
  Measurement points:
  * Distal: at the wrist, 8 cm proximal to the m. abductor pollicis brevis.
  * Proximal: at the cubital fossa
Nerve conduction studies: Motor median nerve proximal latency | 0 and 12 months
  Nerve conduction studies of motor median nerve proximal latency (milliseconds)
  Median nerve measurement points:
  * Distal: at the wrist, 8 cm proximal to the m. abductor pollicis brevis.
  * Proximal: at the cubital fossa
Nerve conduction studies: Motor median nerve amplitude | 0 and 12 months
  Nerve conduction studies of motor median nerve amplitude (millivolts)
  Median nerve measurement points:
  * Distal: at the wrist, 8 cm proximal to the m. abductor pollicis brevis.
  * Proximal: at the cubital fossa
Nerve conduction studies: Motor median nerve conduction velocity | 0 and 12 months
  Nerve conduction studies of motor median nerve amplitude conduction velocity (meters per second)
  Median nerve measurement points:
  * Distal: at the wrist, 8 cm proximal to the m. abductor pollicis brevis.
  * Proximal: at the cubital fossa
Nerve conduction studies: Motor ulnar nerve distal latency | 0 and 12 months
  Nerve conduction studies of motor ulnar nerve distal latency (milliseconds)
  Ulnar nerve measurement points:
  * Distal: at the wrist, 8 cm proximal to the abductor digiti minimi
  * Proximal: 3 cm distal to the medial epicondyle of the elbow
Nerve conduction studies: Motor ulnar nerve proximal latency | 0 and 12 months
  Nerve conduction studies of motor ulnar nerve proximal latency (milliseconds)
  Ulnar nerve measurement points:
  * Distal: at the wrist, 8 cm proximal to the abductor digiti minimi
  * Proximal: 3 cm distal to the medial epicondyle of the elbow
Nerve conduction studies: Motor ulnar nerve amplitude | 0 and 12 months
  Nerve conduction studies of motor ulnar nerve amplitude (millivolts)
  Ulnar nerve measurement points:
  * Distal: at the wrist, 8 cm proximal to the abductor digiti minimi
  * Proximal: 3 cm distal to the medial epicondyle of the elbow
Nerve conduction studies: Motor ulnar nerve conduction velocity | 0 and 12 months
  Nerve conduction studies of motor ulnar nerve conduction velocity (meters per second)
  Ulnar nerve measurement points:
  * Distal: at the wrist, 8 cm proximal to the abductor digiti minimi
  * Proximal: 3 cm distal to the medial epicondyle of the elbow
Nerve conduction studies: Sensory median nerve latency | 0 and 12 months
  Nerve conduction studies of sensory median nerve latency (milliseconds)
  Median nerve measurement points:
  Palmar branch, 8 cm distance, 4th digit with 14 cm distance
Nerve conduction studies: Sensory median nerve amplitude | 0 and 12 months
  Nerve conduction studies of sensory median nerve amplitude (microvolts)
  Median nerve measurement points:
  Palmar branch, 8 cm distance, 4th digit with 14 cm distance
Nerve conduction studies: Sensory median nerve conduction velocity | 0 and 12 months
  Nerve conduction studies of sensory median nerve conduction velocity (meters per second)
  Median nerve measurement points:
  Palmar branch, 8 cm distance, 4th digit with 14 cm distance
Nerve conduction studies: Sensory ulnar nerve latency | 0 and 12 months
  Nerve conduction studies of sensory ulnar nerve latency (milliseconds)
  Ulnar nerve measurement points:
  Palmar branch, 8 cm distance, 4th digit with 14 cm distance
Nerve conduction studies: Sensory ulnar nerve amplitude | 0 and 12 months
  Nerve conduction studies of sensory ulnar nerve amplitude (microvolts)
  Ulnar nerve measurement points:
  Palmar branch, 8 cm distance, 4th digit with 14 cm distance
Nerve conduction studies: Sensory ulnar nerve conduction velocity | 0 and 12 months
  Nerve conduction studies of sensory ulnar nerve conduction velocity (meters per second)
  Ulnar nerve measurement points:
  Palmar branch, 8 cm distance, 4th digit with 14 cm distance
Electromyography: Spontaneous activity | 0 and 12 months
  Electromyography recording spontaneous activity in m.abductor pollicis brevis (Yes/No)
Electromyography: Chronic neurogenic changes | 0 and 12 months
  Electromyography recording chronic neurogenic changes in m.abductor pollicis brevis (Yes/No)
Nerve conduction studies: Bland score | 0 and 12 months
  Scoring of motor and sensory nerve conduction studies using the Bland scoring system (Bland, et al. 2000):
  * 0: normal
  * 1: very mild
  * 2: mild
  * 3: moderate
  * 4: severe
  * 5: very severe
  * 6: extremely severe
  * 7: not gradable
Semmes-Weinstein monofilament test | 0-24 months
  Bilateral test of sensory function in digits 1,2 and 5 using a 2.83 monofilament. Graded absent/present.
Grip strength | 0-24 months
  Test of grip strength using dynamometer. Range 0-90 kg.
Grip ability test (GAT) | 0-24 months
  Simplified version of the Sollerman grip function test. Measures time for subject to perform 3 tasks: Pulling a tubular bandage over the hand, putting a paper clip on an envelope, and pouring water from a jar into a cup. Range 0-60 seconds for each task. Outcome measure is calculated as: tubular bandage (seconds) x 1.8 + paper clip on an envelope (seconds) + pouring water (seconds) x 1.8
Patient assessment of treatment effect on symptoms | 3-24 months
  Patient-reported assessment of treatment effect on symptoms (current state compared to before treatment), reported on a 5-level ordinal (Likert) scale from 1 (best) to 5 (worst).
Patient assessment of expected treatment effect on symptoms | 0 months
  Patient-reported expectation (reported by the patient prior to treatment) of the treatment's effect on symptoms, reported on a 5-level ordinal (Likert) scale from 1 (best) to 5 (worst).
Patient assessment of CTS symptoms | 0-24 months
  Patient-reported assessment of CTS-related symptoms (current state), reported on a 5-level ordinal (Likert) scale from 1 (best) to 5 (worst).
Patient assessment of CTS-related functional impairment | 0-24 months
  Patient-reported assessment of current CTS-related functional impairment (current state), reported on a 5-level ordinal (Likert) scale from 1 (best) to 5 (worst).
Patient assessment of acceptability of CTS-related symptoms and functional disability | 0-24 months
  Patient assessment if the current CTS-related symptoms and functional disability are acceptable (yes or no)
Ultrasound measure of proximal cross-sectional area of the median nerve | 0-24 months
  Bilateral evaluation of the proximal cross-sectional area of the median nerve (square millimeters) (as specified in protocol)
Ultrasound measure of distal cross-sectional area of the median nerve | 0-24 months
  Bilateral evaluation of the distal cross-sectional area of the median nerve (square millimeters) (as specified in protocol)
Ultrasound measures of vascularity of the median nerve in the carpal tunnel | 0-24 months
  Bilateral evaluation of vascularity of the median nerve in the carpal tunnel. Scored 0 to 3
  * 0: no PD signal
  * 1: 1 singular blood vessel
  * 2: 2-3 single blood vessels or 2 confluent
  * 3: ≥4 single blood vessels or ≥ 3 confluent
Disabilities of the Arm, Shoulder, and Hand (Quick-DASH) | 0-24 months
  11-item patient reported outcome measure for disabilities of the arm, shoulder, and hand.
  (Beaton DE, et al. 2005)
Patient pain assessment | 0-24 months
  Patient-reported CTS-related pain on a 0-100 mm visual analogue scale (VAS), where 0 indicates no pain and 100 indicates worst possible pain.
Work Productivity and Activity Impairment Questionnaire (WPAI) | 0-24 months
  Patient-reported outcome of physical function in work and activity. (Reilly MC, et al. 1993)
Days of work absence since start of intervention | 3-24 months
  Number of days of work absence due to CTS or treatment of CTS since start of intervention
EuroQoL 5-dimension health-related quality of life (EQ5D-5L) | 0-24 months
  EuroQoL 5-dimension patient-reported outcome for health-related quality of life.
  (Herdman M, et al. 2011)
Adverse events | 0-24 months
  Number and nature of adverse events and serious adverse events
Successful treatment after 1 corticosteroid injection | 3-24 months
  Only applicable in the injection treatment strategy arm. Subjects who have received 1 corticosteroid injection who have attained a successful treatment result (Boston Carpal Tunnel Questionnaire Symptom Severity Scale ≤ 1.5) without surgery
Successful treatment after 2 corticosteroid injections | 3-24 months
  Only applicable in the injection treatment strategy arm. Subjects who have received 2 corticosteroid injections who have attained a successful treatment result (Boston Carpal Tunnel Questionnaire Symptom Severity Scale ≤ 1.5) without surgery
Successful treatment after secondary surgery | 3-24 months
  Only applicable in the injection treatment strategy arm. Subjects who have received 1 or 2 corticosteroid injections and secondary surgery who have attained a successful treatment result (Boston Carpal Tunnel Questionnaire Symptom Severity Scale ≤ 1.5)
Undergone re-operation | 3-24 months
  Subject have received a re-operation (yes/no)
  A participant who for any reason requires a re-operation, either after primary surgery (surgery arm) or after corticosteroid injection therapy and delayed surgery (injection arm). Reasons for re-operation may, for instance, be wound complications or failure of the initial procedure.
  NOTE: Secondary (delayed) surgery in a participant in the injection arm in accordance with the study treatment algorithm is not considered a re-operation.
Cost of treatment | 0-24 months
  Direct treatment-associated costs, including hospital visits and procedures/interventions. Based on the diagnosis-related group (DRG) pricing system and codified price-lists for medical procedures.

OTHER OUTCOMES:
Use of hospital services | 0-24 months
  Use of hospital services from The Norwegian Patient Register (NPR)
Use of primary care resources | 0-24 months
  Use of primary care resources based on data from Norwegian municipal patient- and user register (KPR)
Work participation | 0-24 months
  Work participation based on data from Statistics Norways's (SSB) event database for social services (FD Trygd)
Total cost | 0-24 months
  Unit costs will be assigned to each type of service by means of the diagnosis-related group (DRG) pricing system, and the price list of the Norwegian Medicines Agency. For each patient total costs will be estimated utilization of health care and social services. The mean symptom severity and cost in the two treatment arms will be used to estimate a cost-effectiveness ratio for the treatment strategies.
Environmental impact analysis | 0-24 months
  Greenhouse gas emissions expressed as CO2 equivalents

CONTACTS AND LOCATIONS:
Overall Officials: Hilde B Hammer, MD, PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (5):
- Norway (5):
  - Akershus University Hospital, Lørenskog, Akershus
  - Department of Surgery and Anesthesiology, Diakonhjemmet Hospital, Oslo, Norge
  - Department of Rheumatology, Diakonhjemmet Hospital, Oslo
  - Department of Orthopedic Surgery, Martina Hansens Hospital, Sandvika
  - Department of Rheumatology, Martina Hansens Hospital, Sandvika

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bland JD. A neurophysiological grading scale for carpal tunnel syndrome. Muscle Nerve. 2000 Aug;23(8):1280-3. doi: 10.1002/1097-4598(200008)23:83.0.co;2-y. PMID 10918269
- [Background] Levine DW, Simmons BP, Koris MJ, Daltroy LH, Hohl GG, Fossel AH, Katz JN. A self-administered questionnaire for the assessment of severity of symptoms and functional status in carpal tunnel syndrome. J Bone Joint Surg Am. 1993 Nov;75(11):1585-92. doi: 10.2106/00004623-199311000-00002. PMID 8245050
- [Background] Beaton DE, Wright JG, Katz JN; Upper Extremity Collaborative Group. Development of the QuickDASH: comparison of three item-reduction approaches. J Bone Joint Surg Am. 2005 May;87(5):1038-46. doi: 10.2106/JBJS.D.02060. PMID 15866967
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777